CLINICAL TRIAL: NCT01486758
Title: Pilot Study: Azithromycin to Prevent Wheezing Following Severe RSV Bronchiolitis
Brief Title: Azithromycin to Prevent Wheezing Following Severe Respiratory Syncytial Virus (RSV) Bronchiolitis
Acronym: APW-RSV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Avraham Beigelman, Assistant Professor of Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201107151; ICTS, Washington University (Other Grant/Funding Number: CTSA402)
Record Dates: First submitted 2011-11-28; First posted 2011-12-06 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: RSV Bronchiolitis
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Active Comparator): Oral azithromycin
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Oral Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Oral azithromycin 10 mg/kg once daily for 7 days followed by 5mg/kg once daily for additional 7 days.
  Arms: Azithromycin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This trial is a proof-of-concept pilot study aim to investigate the biologic and clinical effects of early azithromycin treatment in children hospitalized with Respiratory Syncytial Virus (RSV) bronchiolitis.

HYPOTHESES

In infants hospitalized with RSV bronchiolitis, azithromycin therapy (compared to placebo) will result in:

1. Decreased concentrations of inflammatory mediators (IL-8 as primary outcome) in serum and nasal wash measured on day 8 after randomization.
2. A smaller proportion of participants with recurrent (≥2) wheezing episodes during weeks 3-52 following randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-18 months.
2. Hospitalization for the first episode of RSV bronchiolitis:

   * Confirmed RSV infection by positive nasal swab results (viral culture and/or direct antigen detection) from the SLCH virology lab; AND
   * At least two of the following symptoms/signs of bronchiolitis: respiratory rate greater than 40 breaths/minute; cough; wheezing; audible rales, crackles, and/or rhonchi; paradoxical chest movements (retractions).
3. Duration of respiratory symptoms from initiation of symptoms to admission is 5 days or less. Time of admission will define by the time the child was seen in the ED for the visit that led to hospitalization.
4. Randomization can be performed within 48 hours from time of admission (defined by time of first set of vital signs obtained on the floor).
5. Willingness to provide informed consent by the child's parent or guardian

   -

Exclusion Criteria:

1. Prematurity (gestational age < 36 weeks).
2. Presence or history of other significant disease (CNS, lung, cardiac, renal, GI, hepatic disease, hematologic, endocrine or immune disease). Children with atopic dermatitis will not be excluded from the study.
3. Clinically significant gastroesophageal reflux currently treated with a daily anti-reflux medication (anti- H2 or PPI).
4. The child has significant developmental delay/failure to thrive, defined as weight < 3% for age and gender.
5. History of previous (before the current episode) wheeze or previous treatment with albuterol.
6. Treatment (past of present) with corticosteroid (systemic or inhaled) and/or montelukast.
7. Treatment with any antibiotics in the past 2 weeks.
8. Treatment with Macrolide antibiotic (Azithromycin, clarithromycin or erythromycin) with the past 4 weeks.
9. Current treatment with any daily medication (other then albuterol, vitamins or nutritional supplements).
10. Participation in another clinical trial.
11. Evidence that the family may be unreliable or nonadherent, or may move from the clinical center area before trial completion.
12. Contraindication of use of azithromycin or any other macrolide antibiotics.

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Beigelman, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Department of Pediatrics, Washington University School of Medicine; and St. Louis Children's Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo for 14 days.
Period: Overall Study
Arm/Group | Placebo | Azithromycin
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Azithromycin: Oral azithromycin 10 mg/kg once daily for 7 days followed by 5mg/kg once daily for additional 7 days.
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 9 | 14 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: IL-8 Concentrations
Description: Biological outcome: The difference in IL-8 concentrations, measured in serum on day 8 after randomization, among infants treated with azithromycin and those treated with placebo.
Time Frame: Day 8
Measure: Median (Inter-Quartile Range); unit: Pg/ml
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
Pg/ml | 12,795 [6,265 to 17,763] | 14,676 [7,931 to 19,270]
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; Test type: Superiority or Other; p = 0.6, ANCOVA

2. Primary Outcome: Proportion of Participants Who Experience Subsequent Recurrent (≥2) Wheezing Episodes
Description: Clinical outcome: The difference in the proportion of participants who experience subsequent recurrent (≥2) wheezing episodes among infants treated with azithromycin and those treated with placebo.
Time Frame: 3-52 weeks following randomization
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
Proportion of participants | .50 | .39

3. Secondary Outcome: Concentrations of IL-8 in Nasal Lavage on Day 15
Time Frame: Day 15
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
pg/ml | 2,318 [948 to 5,476] | 865 [357 to 2,212]

4. Secondary Outcome: Rates of Drug Related GI Side Effects.
Time Frame: One month from randomization
Measure: Number; unit: Number of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
Number of participants | 8 | 7

5. Secondary Outcome: Likelihood to Develop 3 or More Wheezing Episodes
Description: Likelihood to develop 3 or more wheezing episodes measured by a Kaplan-Meier survival analysis
Time Frame: Week 3-52
Population: A Kaplan-Meier survival analysis was conducted to compare the likelihood of developing a third episode of wheezing among participants who received azithromycin versus those who received placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
percentage of participants | 50 | 22
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; Test type: Superiority or Other; p = 0.048, Log Rank

6. Secondary Outcome: Respiratory Symptoms Following RSV Bronchiolitis
Description: Number of days with respiratory symptoms (cough, wheeze, or shortness of breath)
Time Frame: 3-52 weeks following randomization
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
Number of days | 70.1 (43.1) | 36.7 (28)

7. Secondary Outcome: Number of Children Who Were Prescribed Inhaled Corticosteroids
Time Frame: 3-52 weeks following randomization
Measure: Number; unit: Number of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
Number of participants | 6 | 1

8. Secondary Outcome: Proportion of Participants With a Physician Diagnosis of Asthma
Description: The proportion of participants with a physician diagnosis of asthma
Time Frame: Week 3-52
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 20 | 19
Percentage of participants | .25 | .11

ADVERSE EVENTS:
Arm/Group | Placebo | Azithromycin
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/19
Other Adverse Events (participants affected / at risk) | 8/20 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Azithromycin (N=19)
Hospitalization for for wheezing episodes (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (3) — 2 participants in the azithromycin group were re-hospitalized for wheezing episodes (3 and 11 months after enrolment) and one patient in the placebo group was hospitalized 3 times for wheezing (all within the first 3 months of the study).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Azithromycin (N=19)
Gastrointestinal adverse events (Gastrointestinal disorders) | 8 (8) | 7 (7) — Gastrointestinal adverse events (diarrhea, vomiting, or abdominal pain) during the treatment phase were recorded in 7 children treated with azithromycin and in 8 children treated with placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes